CLINICAL TRIAL: NCT06114706
Title: Best Assessment of Sore Throat and Antibiotic Prescribing
Acronym: BASTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1299-3543
Record Dates: First submitted 2023-10-23; First posted 2023-11-02 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Pharyngitis
Keywords: Guideline; Sore throat; Pharmacy; Nurses; Physicians
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Intervention Model Description: Parallel groups each with different interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Initial assessement by physicians (Active Comparator): Patients attending with an acute sore throat are initially assessed by a physician. This is one variant of current standard practice.
  Interventions: Behavioral: Physicians assess patients
- Initial assessement by nurses (Active Comparator): Patients attending with an acute sore throat are initially assessed by a nurse. This is one variant of current standard practice.
  Interventions: Behavioral: Nurses assess patients
- Initial assessement by pharmacists (Experimental): Patients attending with an acute sore throat are initially assessed by a pharmacist. This is officially not standard practice in Sweden, although it happens.
  Interventions: Behavioral: Pharmacists assess patients

INTERVENTIONS:
Behavioral: Physicians assess patients — Physicians are asked to assess patients following the current Swedish guideline
  Arms: Initial assessement by physicians
Behavioral: Nurses assess patients — Nurses are asked to assess patients following the current Swedish guideline
  Arms: Initial assessement by nurses
Behavioral: Pharmacists assess patients — Pharmacists are asked to assess patients following the current Swedish guideline
  Arms: Initial assessement by pharmacists

SUMMARY:
This project aims to investigate if an organisational change of patient flow away from medical practitioners can reduce unnecessary antibiotic prescribing in patients attending with a sore throat as the main complaint.

DETAILED DESCRIPTION:
Today patients appear either at a PHC centre or at the Pharmacy. The Pharmacy may provide advice on analgesic or refer the patient to a PHC centre. At the PHC centre, the patient may first appear to the medical practitioner or a nurse pending on local routines. The current Swedish guideline recommends no antibiotics and no testing for patients with 0-2 Centor criteria. For patients with 3-4 Centor criteria the guideline recommends testing and only consider antibiotics if GAS is present.

COVID-19 has gradually transformed from expressing itself as a severe lower respiratory tract infection to be more of an upper respiratory tract infection. Furthermore, COVID-19 is likely to transform from a pandemic to an endemic state with a low continuous incidence. Hence, in response to COVID-19 it seems crucial to identify to what extent the common sore throat is caused by the SARS-CoV-2.

Furthermore, a large controlled clinical trial is required to sort out if patients attending with a sore throat as the main complaint are best managed by medical practitioners, nurses or pharmacists. This study aims to perform such a controlled clinical trial comparing the outcome of sore throat patients management by medical practitioner, nurses and pharmacists. This study also aims to investigate to what extent the SARS-CoV-2 virus is identified in these patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient is contacting/attending PHC centre or Pharmacy presenting with a sore throat as the main complaint.
* Male or female, aged ≥6 years.
* Fluent in Swedish (reading, writing, conversational) (applicable to caregivers/parents/guardians in case of children).
* Mental state such that he or she can understand and give informed consent to participation in the study by signing the Information and Consent Form.
* Provision of signed and dated Informed Consent Form.

Exclusion Criteria:

* The illness episode is classified as potentially complicated or potentially critically ill
* Presence of SARS-CoV-2 virus in a patient first appearing at the PHC in a cluster where the assessment is supposed to be done by the pharmacists. The patient will not be sent to the pharmacist in case of presence of SARS-CoV-2-virus.
* Patient request to be withdrawn from the study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Guideline adherence | Immediately after the consultation
  Will the proportion of patients attending for an uncomplicated acute sore throat being managed according to prevailing guidelines differ if the initial assessment is made by a medical practitioner, a trained nurse or a trained pharmacist

SECONDARY OUTCOMES:
Illness severity | Immediately after the consultation
  What proportion of patients attending PHC centres or pharmacies are classified as apparently uncomplicated, potentially complicated or potentially critically ill
Type of patients seeking care | Immediately after the consultation
  Will patient characteristics differ if the patient first appears to the medical practitioner, a trained nurse or a trained pharmacist?
Presence of SARS-CoV-2 virus | Immediately after the consultation
  To what extent do patients attending Primary Health Care/Pharmacies due to an acute sore throat harbour the SARS-CoV-2 virus?

CONTACTS AND LOCATIONS:
Overall Officials: Ronny Gunnarsson, PhD, Principal Investigator — University of Gothenburg and Region Vastra Gotaland
Locations (4):
- Sweden (4):
  - Apoteket, Stenungsund
  - Närhälsan Stenungsund Vårdcentral, Stenungsund
  - Praktikertjänst Hälsobrunnen Vårdcentral, Ulricehamn
  - Apoteksgruppen, Ulricehamn

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT06114706/Prot_SAP_000.pdf